CLINICAL TRIAL: NCT05010590
Title: Anabolic Therapy in Postmenopausal Osteoporosis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Benjamin Leder, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P002125
Record Dates: First submitted 2021-08-12; First posted 2021-08-18 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-12

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — romosozumab; Denosumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Romosozumab and denosumab (Active Comparator)
  Interventions: Drug: Romosozumab; Drug: Denosumab
- Romosozumab (Active Comparator)
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Romosozumab — Monthly romosozumab
Drug: Denosumab — Every 6 months denosumab
  Arms: Romosozumab and denosumab

SUMMARY:
In this research study we want to learn more about the effect of two different FDA-approved medications in the treatment of osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women at high risk of fracture

Exclusion Criteria:

* Prior therapy exclusions

  1. current use or use in the past 12 months of oral bisphosphonates or denosumab
  2. current use or use within the past 3 months of estrogens, SERMs, or calcitonin.
  3. use of oral or parenteral glucocorticoids for more than 14 days within the past 6 months
  4. any current or previous use of romosozumab or strontium
  5. current use or use within the past 3 years of teriparatide, abaloparatide, or any parenteral bisphosphonate.

Other exclusions

1. Confirmed serum alkaline greater than 2 times the upper normal limit.
2. Stage 4 or 5 chronic kidney disease (GFR less than 30)
3. Hypercalcemia (Ca greater than 10.5 mg/dL)
4. Hypocalcemia (Ca less than 8.8 mg/dL)
5. Elevated blood PTH (intact PTH greater than 77 pg/mL)
6. Serum 25-OH vitamin D less than 20 ng/mL
7. HCT less than 32%.
8. History of malignancy (except basal cell carcinoma).
9. Significant pulmonary disease
10. History of myocardial infarction or stroke within the preceding year.
11. History of unstable angina or transient ischemic attack in the past year.
12. Current atrial fibrillation.
13. Any health condition that, in the opinion of the study physician, significantly increases the risk of cardiovascular events.
14. Major psychiatric disease that in the opinion of the investigator would preclude the subject from providing adequate informed consent or completing the protocol procedures.
15. Excessive alcohol use or substance abuse that in the opinion of the investigator would preclude the subject from providing adequate informed consent or completing the protocol procedures.
16. Uncontrolled eczema
17. Congenital or acquired bone disease other than osteoporosis.
18. Known sensitivity to denosumab or any of its excipients.
19. Known sensitivity to romosozumab or any of its excipients.
20. History of osteonecrosis of the jaw, extensive dental work involving extraction or dental implants in the past 3 months, or extensive dental work planned in the upcoming 12 months.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 50 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Total hip areal bone mineral density | Month 0 to 12
  Change in total hip bone density between month 0 and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Leder, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leder BZ, Ramchand SK, Jordan M, Ryan S, Patnaik A, Lee H, Tsai JN. 3 months vs 12 months of romosozumab for postmenopausal osteoporosis (LIDA): an open-label, non-inferiority, randomised controlled trial. Lancet Diabetes Endocrinol. 2026 Jan 29:S2213-8587(25)00319-5. doi: 10.1016/S2213-8587(25)00319-5. Online ahead of print. PMID 41621431